CLINICAL TRIAL: NCT04781751
Title: Ultrasonographic Insulin Versus Dexamethasone Injection With Local Anestheticss in Diabetic Patients With Mild to Moderate Median Nerve Entrapement Neuropathy .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 212/2-2021
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Pain, Neuropathic
MeSH Terms: conditions — Neuralgia | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexamethasone (No Intervention): dexamethasone with local anesthetics injected for carpal tunnel relief
- Insulin group (Active Comparator): insulin with local anesthetics and dexamehtasone injected for carpal tunnel relief
  Interventions: Drug: insulin injection

INTERVENTIONS:
Drug: insulin injection — Carpal tunnel syndrome sonagraphic injection
  Arms: Insulin group

SUMMARY:
Insulin injection in carpal tunnel compared with dexamethsone in diabetic patients

DETAILED DESCRIPTION:
Trial to decrease median nerve entrapement neuropathy recurrence using insulin co-injection

ELIGIBILITY:
Inclusion Criteria:

* All diabetic patients with carpal tunnel syndrome

Exclusion Criteria:

* Refusal to participate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-04-05 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
pain relief | 12 weeks
  consumption analgesics

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, ALMinya, Egypt